CLINICAL TRIAL: NCT03294759
Title: Pilot Study: Augmentation of ACL Reconstruction With Bone Marrow Stem Cells and Amnion Collagen Matrix Wrap
Brief Title: Bio ACL Reconstruction Amnion Collagen Matrix Wrap and Stem Cells
Acronym: BioACLRCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio ACL (RCT)
Record Dates: First submitted 2017-09-20; First posted 2017-09-27 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
Keywords: amion; stem cell; acl
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — cancer procoagulant

STUDY DESIGN:
Intervention Model Description: ACL harvested for autograft reconstruction of the ACL with either hamstring or patellar tendon grafts. The graft will be wrapped in a collagen wrap and injection with aspirate from the patient's bone marrow.
  The control group will have standard ACL reconstruction with either hamstring or patellar tendon grafts.
Who Masked: Participant, Outcomes Assessor
Masking Description: Bone marrow aspirate will be collected through the surgical site from the distal femur with a trocar designed for this purpose. Therefore patients will be unable to determine if they have had stem cells harvested
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bio-ACL (Amion) (Experimental): Intervention: ACL Autograft Reconstruction with Amion Collagen Scaffold. Stem Cells isolated from bone marrow aspirate from distal femur will be injected inside the Amion Collagen Scaffold.
  Interventions: Other: Bio ACL
- Control (Active Comparator): Intervention: Normal ACL Autograft Reconstruction with either patella or hamstring autograft will be performed in the control group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Bio ACL — Bone marrow aspirate will be centrifuged using the Arthrex Angel system to optimally concentrate the cells for implantation. The graft for the experimental groups will be wrapped with a sterile amnion matrix wrap, supplied by Arthrex
  Other Names: Amnion
  Arms: Bio-ACL (Amion)
Other: Control — Normal ACL reconstruction technique with either patella or hamstring autograft
  Other Names: Standard ACLr
  Arms: Control

SUMMARY:
Collagen based -membrane derived from amniotic tissue can be used to help reestablish the natural synovial lining of the reconstructed ACL, in effect acting as both a barrier from the synovial fluid and as a scaffold to contain autologous mesenchymal stem cells and growth factors contiguous with the graft, thus aiding and perhaps accelerating the natural maturation and ligamentization process of the implanted graft tissue. Acceleration and improvement in graft maturation and strength would be a significant advancement in sports medicine allowing safer and earlier return to sports and activity

DETAILED DESCRIPTION:
Histologic studies have determined that graft ligamentization following anterior cruciate ligament (ACL) reconstruction may take from 6 to 18 months. (1) It has been reported that incomplete graft maturation and incorporation is one cause of clinical graft failure. Animal studies have illustrated improved tendon healing/integration in ACL models augmented with stem cell technologies. (2-4). Basic scientists theorize that optimization of stem cell treatments for tissue regeneration requires that a "regenerative triad" be employed, i.e., use of a scaffold, stem cells and growth factors. In the intra-articular environment, research has shown that a scaffold such as an amnion wrap is necessary to contain the stem cells and growth factors in close proximity to the ACL graft. (2, 4, 5)

The normal, uninjured human ACL is covered by a layer of synovial tissue which contributes to the blood supply and nutrition of the native ACL. It is theorized that the lack of a synovial lining after injury and following traditional ACL reconstruction contributes to slow ligamentization and possible failure of reconstructed grafts.(5) Two studies have demonstrated accelerated maturation and ligamentization of human ACL graft augmented with point of care blood products. (6, 7) In one, leucocyte poor platelet rich plasma was injected directly into the body of the graft. (6) In the other, the platelet derived growth factors were loaded in a gelatin carrier which was wrapped around the graft. (7) In both studies accelerated and increased ligament maturation was documented compared to the controls. Collagen membranes derived from amniotic tissue have been successful to aid healing when used in difficult wounds and meniscal repair surgery. (8, 9)

The use of a collagen based -membrane derived from amniotic tissue may be used to help reestablish the natural synovial lining of the reconstructed ACL, in effect acting as both a barrier from the synovial fluid and as a scaffold to contain autologous mesenchymal stem cells and growth factors contiguous with the graft. Thus aiding and perhaps accelerating the natural maturation and ligamentization process of the implanted graft tissue. Acceleration and improvement in graft maturation and strength would be a significant advancement in sports medicine allowing safer and earlier return to sports and activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 45 who are scheduled to have anterior cruciate ligament reconstruction with autologous grafts by one of the investigating physicians will be screened for participation in this study.
* Patients must be willing to undergo MRI scans post -operatively at 3, 6, 9 months and 1 year

Exclusion Criteria:

* Patients with prior procedures or significant prior injuries to the same knee are excluded. - - Any patient who will have difficulty obtaining internet access, does not have an active e-mail address, or is unable to comprehend study documents or give informed consent will be excluded.
* Patient who are unable to complete MRI examinations due to claustrophobia or anxiety will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
Changes in ACL | 3 months, 6 months, 9 months, 12 months post-op
  MRI region of interest mapping to produce mean T2 values

SECONDARY OUTCOMES:
Changes in patient-reported pain rating | 3 months, 6 months, 9 months, 12 months post-op
  Visual analog scale will be used to assess pain
Changes in Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 months, 6 months, 9 months, 12 months post-op
  Patients will complete KOOS questionnaire on SOS
Changes in Short Form 12 (SF-12) patient ratings | 3 months, 6 months, 9 months, 12 months post-op
  Patients will complete SF-12 questionnaire on SOS
Changes in Single Assessment Numerical Evaluation (SANE) patient ratings for function | 3 months, 6 months, 9 months, 12 months post-op
  Patients will complete the SANE questionnaire on SOS
Marx Activity Scale Rating | 12 months post-op
  Patients will complete the Marx Activity questionnaire on SOS

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, MD, Principal Investigator — Andrews Research & Education Foundation
Locations (1):
- Andrews Institute, Gulf Breeze, Florida, United States

REFERENCES:
- [Background] Claes S, Verdonk P, Forsyth R, Bellemans J. The "ligamentization" process in anterior cruciate ligament reconstruction: what happens to the human graft? A systematic review of the literature. Am J Sports Med. 2011 Nov;39(11):2476-83. doi: 10.1177/0363546511402662. Epub 2011 Apr 22. PMID 21515806
- [Background] Matsumoto T, Kubo S, Sasaki K, Kawakami Y, Oka S, Sasaki H, Takayama K, Tei K, Matsushita T, Mifune Y, Kurosaka M, Kuroda R. Acceleration of tendon-bone healing of anterior cruciate ligament graft using autologous ruptured tissue. Am J Sports Med. 2012 Jun;40(6):1296-302. doi: 10.1177/0363546512439026. Epub 2012 Mar 16. PMID 22427618
- [Background] Mifune Y, Matsumoto T, Takayama K, Terada S, Sekiya N, Kuroda R, Kurosaka M, Fu FH, Huard J. Tendon graft revitalization using adult anterior cruciate ligament (ACL)-derived CD34+ cell sheets for ACL reconstruction. Biomaterials. 2013 Jul;34(22):5476-87. doi: 10.1016/j.biomaterials.2013.04.013. Epub 2013 Apr 28. PMID 23632324
- [Background] Joshi SM, Mastrangelo AN, Magarian EM, Fleming BC, Murray MM. Collagen-platelet composite enhances biomechanical and histologic healing of the porcine anterior cruciate ligament. Am J Sports Med. 2009 Dec;37(12):2401-10. doi: 10.1177/0363546509339915. PMID 19940313
- [Background] Sanchez M, Anitua E, Azofra J, Prado R, Muruzabal F, Andia I. Ligamentization of tendon grafts treated with an endogenous preparation rich in growth factors: gross morphology and histology. Arthroscopy. 2010 Apr;26(4):470-80. doi: 10.1016/j.arthro.2009.08.019. Epub 2010 Jan 15. PMID 20362825
- [Background] Radice F, Yanez R, Gutierrez V, Rosales J, Pinedo M, Coda S. Comparison of magnetic resonance imaging findings in anterior cruciate ligament grafts with and without autologous platelet-derived growth factors. Arthroscopy. 2010 Jan;26(1):50-7. doi: 10.1016/j.arthro.2009.06.030. PMID 20117627
- [Background] DiDomenico LA, Orgill DP, Galiano RD, Serena TE, Carter MJ, Kaufman JP, Young NJ, Zelen CM. Aseptically Processed Placental Membrane Improves Healing of Diabetic Foot Ulcerations: Prospective, Randomized Clinical Trial. Plast Reconstr Surg Glob Open. 2016 Oct 12;4(10):e1095. doi: 10.1097/GOX.0000000000001095. eCollection 2016 Oct. PMID 27826487
- [Background] Piontek T, Ciemniewska-Gorzela K, Naczk J, Jakob R, Szulc A, Grygorowicz M, Slomczykowski M. Complex Meniscus Tears Treated with Collagen Matrix Wrapping and Bone Marrow Blood Injection: A 2-Year Clinical Follow-Up. Cartilage. 2016 Apr;7(2):123-39. doi: 10.1177/1947603515608988. Epub 2015 Nov 30. PMID 27047635
- [Background] Li H, Tao H, Cho S, Chen S, Yao Z, Chen S. Difference in graft maturity of the reconstructed anterior cruciate ligament 2 years postoperatively: a comparison between autografts and allografts in young men using clinical and 3.0-T magnetic resonance imaging evaluation. Am J Sports Med. 2012 Jul;40(7):1519-26. doi: 10.1177/0363546512443050. Epub 2012 Apr 11. PMID 22495290
- [Background] Biercevicz AM, Akelman MR, Fadale PD, Hulstyn MJ, Shalvoy RM, Badger GJ, Tung GA, Oksendahl HL, Fleming BC. MRI volume and signal intensity of ACL graft predict clinical, functional, and patient-oriented outcome measures after ACL reconstruction. Am J Sports Med. 2015 Mar;43(3):693-9. doi: 10.1177/0363546514561435. Epub 2014 Dec 24. PMID 25540298
- [Background] Riboh JC, Saltzman BM, Yanke AB, Cole BJ. Human Amniotic Membrane-Derived Products in Sports Medicine: Basic Science, Early Results, and Potential Clinical Applications. Am J Sports Med. 2016 Sep;44(9):2425-34. doi: 10.1177/0363546515612750. Epub 2015 Nov 19. PMID 26585668
- [Background] Baeten D, Van den Bosch F, Elewaut D, Stuer A, Veys EM, De Keyser F. Needle arthroscopy of the knee with synovial biopsy sampling: technical experience in 150 patients. Clin Rheumatol. 1999;18(6):434-41. doi: 10.1007/s100670050134. PMID 10638766
- [Derived] Anz AW, Jordan SE, Ostrander RV 3rd, Branch EA, Denney TS, Cohen A, Andrews JR. Augmentation of ACL Autograft Reconstruction With an Amnion Collagen Matrix Wrap and Bone Marrow Aspirate Concentrate: A Pilot Randomized Controlled Trial With 2-Year Follow-up. Orthop J Sports Med. 2023 Nov 17;11(11):23259671231210035. doi: 10.1177/23259671231210035. eCollection 2023 Nov. PMID 38021297

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT03294759/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03294759/ICF_001.pdf